CLINICAL TRIAL: NCT00528762
Title: Mexican and African American Family Focus Groups on Puberty
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2006-0113
Record Dates: First submitted 2007-09-11; First posted 2007-09-12 (Estimated); Last update posted 2012-07-30 (Estimated); Status verified 2012-07

CONDITIONS: Healthy
Keywords: Epidemiology; Puberty; Body Weight; Body Image; Focus Group
MeSH Terms: conditions — Body Weight | interventions — Focus Groups

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Focus Group: Mexican American or African American females (aged 6-12 years old) and their parents
  Interventions: Behavioral: Focus Group

INTERVENTIONS:
Behavioral: Focus Group — Focus group discussion about puberty and body image lasting 1 1/2 hours.

SUMMARY:
Primary Objective:

For focus groups of Mexican American and African-American girls and focus groups of their parents to explore factors that could enhance the conduct of a future study of puberty and body mass.

Specifically these focus groups will address:

* Whether clinical assessment of pubertal staging is acceptable.
* How to enhance cooperation by parents and their daughters of different socioeconomic groups, among families with different levels of acculturation, and girls of different body mass indices.
* Explore whether established questionnaire items about puberty, that have been used in traditional surveys, require culture-specific changes to improve exposure assessment.
* Explore the acceptability of self-reported pictograms for body image and for developmental assessment by girls.

DETAILED DESCRIPTION:
For Parents:

This study will involve 5 focus groups. Mothers will take part in 1 of 2 focus groups with other mothers. Fathers will take part in a focus group with other fathers. Girls will take part in 1 of 2 focus groups with other girls. Any eligible parent will be able to participate even if the daughter chooses not to participate in the focus group activities. At the start of each focus group, the moderators will begin with a general session about health related topics, but for the girls, any discussion about pubertal development will take place in two separate groups, with the 6-9 yr olds in one group and 10-12 yr olds in another group. Each group will have about 8 to 10 participants who are all comfortable speaking the same language.

The focus groups will be led by a moderator, a person who will lead the talk and answer any questions participants may have. The moderator will speak both English and Spanish, and you will be assigned to the group where your preferred language is spoken. The discussions will involve talk about puberty and body image, such as the typical age for a girl to start puberty, body changes girls go through in puberty, and girls' level of comfort with how their body looks. Parents of the girls will also be asked to compare their experiences during puberty with their daughters' experiences.

Researchers want to know if you would be comfortable with your daughter taking part in a clinical research study that is planned for the future. Information about this future study will also be presented to each group for discussion. The focus group talks will last about 1 1/2 hours. They will be conducted in the community where you live. You will be told the location before you agree to take part in this study.

All of the discussions will be audio taped and will be kept confidential. The tapes will not be heard by anyone other than the research staff. They will be kept safe in a locked cabinet that stores other confidential research materials, and will be destroyed at the end of this study.

Your participation in this study will be over after your focus group discussion has ended.

This is an investigational study. Up to 50 parents will take part in this study. All will be enrolled at M. D. Anderson.

For Children:

This study will have 5 focus groups per ethnic groups. Mothers will be in 1 of 2 focus groups with other mothers. Fathers will be in a focus group with other fathers. The moderator will speak both English and Spanish, and you will be assigned to the group where your preferred language is spoken. Girls will be in 1 of 2 focus groups with other girls. At the start of each focus group, the moderators will begin with a general session about health related topics, but for the girls, any discussion about pubertal development will take place in two separate groups, with the 6-9 yr olds in one group and 10-12 yr olds in another group. Each group will have about 8 to 10 participants who are all comfortable speaking the same language.

The focus groups will be led by a moderator, a person who will lead the talk and answer any questions participants may have. The discussions will involve talk about your thoughts on growth and development and body image, such as the age you started developing, how your body changes, and your level of comfort with how your body looks. Your parent(s) will also be asked to compare their experiences during puberty with your experience. You will also be asked about your level of comfort with a visit to the doctor and with having your blood drawn and needle sticks.

Researchers also want to know if you would be comfortable taking part in a clinical research study that is planned for the future. Information about this future study will also be presented to each group for discussion. The focus group talks will last about 1 1/2 hours.

All of the discussions will be audio taped and will be kept confidential. The tapes will not be heard by anyone other than the research staff. They will be kept safe in a locked cabinet that stores other confidential research materials, and will be destroyed at the end of this study.

Your participation in this study will be over after your focus group discussion has ended.

This is an investigational study. You will be given the art projects that you created during your focus group for your time and participation. Up to 50 girls will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Mexican American Daughters Inclusion Criteria: must be Mexican or of Mexican-American descent, girls must be aged 6-12 at the time they are contacted to participate in the focus groups. They must be able to communicate in a group in either English or Spanish, must be able to attend the focus group and have a mother who is willing to participate. They must live in a household where there is at least 1 adult participating in the Mano a Mano Cohort study (CPN00-367)
2. African American Daughters Inclusion Criteria: must be African-American descent, girls must be aged 6-12 at the time they are contacted to participate in the focus groups. They must be able to communicate in a group in English, must be able to attend the focus group and have a mother who is willing to participate.
3. Mexican American Mothers Inclusion Criteria: Mothers must be Mexican or of Mexican-American descent, should have a daughter aged 6-12 (index child) at the time they are contacted to participate in the focus groups. They must willing to participate and must live in the same household as the index child at least 5 or more days per week. They must be able to communicate in a group in either English or Spanish and must live in a household where there is at least 1 adult participating in the Mano a Mano Cohort study (CPN00-367)
4. African American Mothers Inclusion Criteria: Mothers must be African-American descent, should have a daughter aged 6-12 (index child) at the time they are contacted to participate in the focus groups. They must willing to participate and must live in the same household as the index child at least 5 or more days per week. They must be able to communicate in a group in English.
5. Mexican American Fathers Inclusion Criteria: Fathers must be Mexican or of Mexican-descent, have a daughter aged 6-12 (index child) at the time they are contacted to participate in the focus groups. They must be willing to participate, live in the same household as the index child at least 5 or more days per week, must be able to communicate in a group in either English or Spanish, and they must live in a household where there is at least 1 adult participating in the Mano a Mano Cohort study (CPN00-367)
6. African American Fathers Inclusion Criteria: Fathers must be African-American descent, have a daughter aged 6-12 (index child) at the time they are contacted to participate in the focus groups. They must be willing to participate, live in the same household as the index child at least 5 or more days per week, must be able to communicate in a group in English.

Exclusion Criteria:

1. Mothers Exclusion Criteria: Mothers will be excluded from the focus group if they are a current MDACC employee, have recently participated in other focus groups or research discussions.
2. Fathers Exclusion Criteria: Fathers will be excluded if they are a current MDACC employee, have recently participated in other focus groups or research discussions.

Ages: 6 Years to 12 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Participants are females aged 6-12 years old that are of Mexican American or African American descent and their parents.
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2006-11; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Exploratory Results from Mexican and African American Family Focus Groups on Puberty | 2 Years

CONTACTS AND LOCATIONS:
Overall Officials: Michele Forman, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- U.T. M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org